CLINICAL TRIAL: NCT02457637
Title: Chinese Chronic Liver Failure Consortium Acute-on-Chronic Liver Disease and Failure Study --a Prospective Multi-center Study in China, the Largest Hepatitis B Virus High-endemic Region.
Brief Title: Chinese CLIF-C Acute-on-Chronic Liver Disease and Liver Failure Study
Acronym: Ch-CANONIC
Status: Completed | Type: Observational
Sponsor: Hai Li (Other)
Responsible Party: Sponsor-Investigator, Hai Li, Professor, Department of Gastroenterology, RenJi Hospital ; Vice Director of the National Digestive Key Laboratory; Youth Commission of Chinese Society of Hepatology., Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: CHINA-ACLF
Record Dates: First submitted 2015-01-31; First posted 2015-05-29 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Liver Failure, Acute on Chronic
Keywords: acute-on-chronic liver disease; acute decompensation; multiple organ failures; acute on chronic liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, stool, liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute-on-Chronic Liver Disease Inpatient: 1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients; and non-alcoholic fatty liver disease patients.
  2. ALI(acute liver injury): including [ALT>3NL(normal level),AST>3NL or TB>2NL within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy, bacterial infection gastrointestinal bleeding or jaundice(TB>5NL)within 1 month before enrollment)].
  3. Standary therapy
  Interventions: Other: Standary therapy

INTERVENTIONS:
Other: Standary therapy — Standary therapy for chronic liver disease with ALI and/or AD

SUMMARY:
Acute on chronic liver failure (ACLF) is a distinct entity encompassing the acute deterioration of liver function, culminating in multiple organs failure and high short-term mortality. Currently, there are differences in definitions and descriptions between western and eastern types of ACLF, especially in the definition of chronic liver disease and its precipitating events. The CANONIC (EASL-CLIF ACLF in Cirrhosis) study put forward CLIF-SOFA (chronic liver failure-sequential organ failure assessment) scores as the clinical diagnostic criteria of ACLF in 2013. Although the Asian Pacific Association for the Study of the Liver (APASL) reached a consensus for diagnostic criteria of ACLF in 2008, it is based on expert opinion. This prospective multicenter clinical trial is launched to clarify the eastern type of ACLF (HBV related) and estimate whether the eastern and western (alcoholic related) types are homogenous. 3 key points of concern are: (1) Whether HBV and non-HBV ACLFs are belonged to a homogenous disease entity which share the same diagnostic criteria, disease grades classification and prognostic model? (2) Whether acute deteriorating patients from cirrhosis or from mild fibrosis (S1-S2) belong to a homogenous entity? (3) To clarify if there are heterogenous groups in APASL criteria diagnosed ACLF patients.

14 Chinese national wide liver centers have been included. Continuous hospitalized chronic liver disease patients of various etiologies (including both cirrhotic and non-cirrhotic) with acute decompensation (AD) or acute hepatic injury (ALI) (aminotransferase > 3NL(normal level)) will be recruited from January to December 2015. Biochemical parameters, organ failure will be collected and evaluated at day 1,4,7,14,21 and 28 after enrollment. Patients'death and LT (liver transplantation) are the primary and secondary endpoints of observation. Mortality and LT rate will be calculated at 28 days,90 days,180 days,1 year and 2 years after enrollment. Considering there will lack of liver biopsy in most of the patients, both CT and FibroScan as supplementary methods to differentiate non-cirrhotic patients. The patients will be continuously followed up once a month until the 24th month after hospital discharging and follow similar hospitalization process again whenever they have new ALI or AD. Data about the patients from stable chronic liver disease to deterioration will be acquired analyzed according to the questions hoped to resolve.

DETAILED DESCRIPTION:
Acute-on chronic liver failure (ACLF) was first described by Japanese researchers in 1995. In 2011, the American Association for the Study of Liver Disease (AASLD) and the European Association for the Study of the Liver (EASL) concluded that the core characteristics of ACLF were multiple organ failures and high short-term mortality. In 2013, the EASL-CLIF (the European Association for the Study of The Liver-chronic liver failure) established the CLIF-SOFA (chronic liver failure-sequential organ failure assessment) criteria of ACLF through a prospective multicenter study at 29 liver units in eight European countries for 1 year, with a focus on patients with alcoholic cirrhosis with acute decompensation (AD). In China, patients with acute deterioration of previously chronic liver disease were diagnosed with chronic severe hepatitis, until 2008 these patients had been termed "ACLF", due to the APASL reached a consensus of diagnostic criteria of ACLF. In the Asia-Pacific region, the majority of liver disease is viral hepatitis, while in western countries, it is alcoholic liver disease. There is a sharp east-west divide with respect to the definition of ACLF, especially in the definition of chronic liver disease and its precipitating events.

The investigators analyzed 6 years' data of hepatitis B virus (HBV)-related chronic liver disease in patients with AD in two affiliated hospitals of Shanghai Jiao Tong University School of Medicine. These data were also quantified and sent to the EASL-CLIF centre for analysis. 80% of whole patients were clinically diagnosed with cirrhosis, 30% of which had pathological diagnosis. Through analysis of the liver tissues of the liver transplantation (LT) patients, 95% had pseudolobules. The residual 5% of liver tissues were in the S3 stage of progressive liver fibrosis. Compared with the CANONIC (EASL-CLIF Acute-on-Chronic Liver Failure in Cirrhosis), there are many similarities between ACLF patients with alcoholic cirrhosis or HBV induced cirrhosis: (1)The age of ACLF patients is younger than that of cirrhotic patients with AD. (2)ACLF is exist at any stage of liver fibrosis. (3)The number of organ failures decides the severity of the disease and is related to mortality of the patient. (4) Predisposition to acute liver injury (ALI) does not correlate with the history of the disease and outcome of the patient. (5)The 90-day mortality rate of ACLF is 45-50%, which is obviously higher than that of non-ACLF patients (5%). (6)Eastern and western types of ACLF can have similar SOFA scores as a diagnostic criterion (CLIF-OF or CLIF-SOFA), and a similar prognostic model to predict the outcomes of ACLF and non-ACLF patients. ACLF patients with cirrhosis induced by HBV or alcoholism differ in main types of organ failure. The former group is liver failure (total bilirubin≥12mg/dl) and coagulation failure(international normalized ratio; INR≥2.5), whereas the latter group is renal failure(creatinine≥2mg/dl or use of renal replacement therapy) and nervous system failure(hepatic encephalopathy; HE≥III grade).

Research on hepatic pathology in HBV-induced ACLF patients after LT in RenJi Hospital demonstrated that the pathological characteristics of ACLF may be MHN/SMHN (massive hepatic necrosis/submassive hepatic necrosis) in the background of liver pseudolobules. Regeneration of hepatic progenitor cells, cholestasis, and sepsis are other possible pathological features of ACLF.

It is necessary to conduct a prospective multicentre study to clarify the eastern type of ACLF and the differences between the eastern and western types of ACLF. The investigators are going to identify three key points: (1)Whether HBV and non-HBV ACLFs are belong to a homogenous disease entity which share the same diagnostic criteria, disease grades classification and prognostic model; (2) Whether acute deteriorating patients from cirrhosis or from mild fibrosis (S1-S2) belong to a homogenous entity? (3)To clarify if there are heterogenous groups in APASL criteria diagnosed ACLF patients.

The investigators plan to enroll 2000-3000 consecutive patients from January to December 2015. The research will be carried out in about 14 Chinese national wide liver centers each of whose total beds are around 500.

The research has two stages. The first stage will be enrollment of 2000-3000 consecutive patients from January to December 2015. Only chronic liver disease patients of various etiologies with AD or ALI will be enrolled. Biochemical parameters, organ failure evaluation, imaging test results treatment therapies will be recorded at day 1,4,7,14,21 and 28 (or last visit date) after enrollment according to case report form. If the patients die or undergo LT, the data at the 24h prior to death or LT will be also recorded. The second stage will be follow-up from January 2016 to December 2017. If the patients improve and are discharged, 24 months' follow-up should be conducted. Whenever the patients die or have LT, the study will be end. Follow-up will be clinical visiting, but telephone call will be acceptable for patients unable to attend. During follow-up, patients will be hospitalized again whenever they have new ALI or AD. Similar data will be collected reference to their prior admission and follow-up will restart.

Every patient will have a unique number. As soon as they are hospitalized, name, age, sex, ID(identification) number, telephone number, e-mail address, WeChat(a popular mobile phone text and voice messaging communication service) number, family address, and degree of education will be collected. The investigators will get the history and etiology of their liver disease, such as hepatitis B, alcoholic liver disease, and autoimmune liver disease. For viral hepatitis, the investigators will ask how antiviral therapy is conducted. The investigators will ascertain if the patients have a history of cirrhosis and for how long. The investigators will ascertain if the patients have any of the following predisposing factors: HBV reactivation, bacterial infection, active alcohol intake, HBV superimposed by other hepatitis viruses, gastrointestinal bleeding, portal vein thrombosis, surgery, intake of hepatotoxic drugs or herbs, or physiological exhaustion. The investigators will establish the main cause of admission: gastrointestinal bleeding, hepatic encephalopathy, ascites, bacterial infection or ALI. The investigators will determine whether the patients have chronic disease such as hypertension, coronary heart disease, diabetes, chronic renal disease, or connective tissue disease.

During hospitalization, data will be collected at 1, 4, 7,14, 21 and 28 days (or last visit date, if the patient is hospitalized less than 28 days), and 24h prior to death or LT (if the patient dies or has LT) and focus on the following three aspects.

The first aspect is evaluation of organ failure. The circulatory system will be evaluated by measuring heart rate and blood pressure and use of vasopressors. Renal function will be evaluated by serum creatinine or renal replacement therapy. Coagulation function will be evaluated by INR (international normalized ratio of prothrombin time). Liver function will be evaluated by serum total bilirubin. The respiratory system will be evaluated by the ratio of oxyhemoglobin saturation and fraction of inspired oxygen. The nervous system will be evaluated by the grade of hepatic encephalopathy. Bacterial infection, including pneumonia, urinary tract infection, spontaneous bacterial peritonitis, spontaneous bacteremia, and cellulitis will be evaluated by positive culture results or imaging findings. Systemic inflammatory reactive syndrome, sepsis, severe sepsis and septic shock will also be assessed. Gastrointestinal bleeding before and after admission, treatment with diuretics, and paracentesis will be recorded. The investigators will establish whether ascites and hepatic encephalopathy can be medically controlled.

The second aspect is laboratory examinations. Tests at admission will include routine blood, urine and stool tests, liver and renal function tests, blood electrolytes, blood-gas analysis, blood glucose, coagulation test, C-reactive protein (CRP), procalcitonin (PCT), HBV antibodies and antigens, anti-hepatitis A (IgM), HBV-DNA, anti-hepatitis E (IgM), anti-hepatitis C, and immunoglobulins (IgA, IgG, IgM and IgM-4). Tests at other times will include blood, urine and stool routine tests, liver and renal function tests, blood electrolytes, blood glucose, coagulation test, CRP and PCT (procalcitonin). Tests optionally done during hospitalization will include autoantibody measurement, blood culture(if the patients have fever and shivering), sputum culture(if there is suspicion of pulmonary infection),middle urine cultivation(when there is suspicion of urinary tract infection) and ascites culture(when there is suspicion of spontaneous bacterial peritonitis).

The third aspect is imaging. During hospitalization, thoracic X ray or computed tomography (CT) will be done to diagnose pulmonary infection. Abdominal CT (enhanced when necessary), B ultrasound and FibroScan or other elastography will be done to diagnose cirrhosis (or fibrosis), portal thrombosis, esophageal and gastric varices and hepatocellular carcinoma.

Patients will be followed up regularly after discharge. When the patients die during follow-up, the time of death and main cause of death will be noted. When the patients undergo LT during follow-up, the time of LT and the results of hepatic pathology will be noted.

Follow-up is by clinical visiting or telephone call depending on whether the patient can attend the clinic. Clinical follow-up is once a month for 2 years adding to 24 visits. The time of visit will be recorded. Antiviral therapy and alcohol intake will be monitored(if the patient has). Laboratory tests include routine blood tests, liver and renal function test, coagulation test, CRP and PCT. B ultrasound will be done to monitor cirrhosis (or fibrosis) and hepatocellular carcinoma. Telephone follow-up will be at 28 days, 3, 6,9, 12, 15, 18, 21 and 24 months. The investigators will determine whether there are new complications (e.g. gastrointestinal bleeding, hepatic encephalopathy, ascites, bacterial infection) and hepatocellular carcinoma.

Referring to the structure of the clinical research of CANONIC study, the investigators will meet every three months to exchange results and ideas. All young committee members from Chinese Society of Hepatology can campaign for joining in this research. There will be a core group with 3-4 members comprising experts with an interest in ACLF. These core members will be responsible for making policies. Members of core group are flexible. Monopolizing and arbitrariness should be forbidden.

Independent departments of gastroenterology, hepatology or infectious diseases are a requirement of the hospitals. Every hospital should have only one principal investigator (PI) as their representative. The PI should be the head of the department and involved in clinical work. The PI should make ward rounds at least twice weekly and evaluate the patients beside the bed. Young members of Chinese Society of Hepatology will be prioritized for the PI. If the young members do not undertake clinical work, they can recommend an eligible attending physician.

There are some measures to guarantee the quality of follow-up. First, set up fast-track follow-up cards for each patient. These patients have priority to make an appointment and see a doctor. Second, every PI should have their assistants. Every assistant is equipped with a cellphone so that patients can call to visit a doctor immediately or be hospitalized in an emergency. Third, set up a WeChat group for patients to inform them about follow-up 1 week in advance. Fourth, every assistant should master the follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

* inpatient (hospitalization >1 days)(including patient in emergency observation wards)
* chronic liver disease patients including non-alcoholic fatty liver disease patients,chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients and decompensated cirrhosis patients
* having acute liver injury [ALT(alanine aminotransferase)>3NL(normal level),AST(aspartate aminotransferase)>3NL or TB(total bilirubin)>2NL within 1 week before enrollment] or acute decompensation[having ascites, hepatic encephalopathy, bacterial infection ,gastrointestinal bleeding or jaundice(TB>5NL)within 1 month].

Exclusion Criteria:

* pregnancy
* hepatocellular carcinoma or other liver malignancies
* malignancy of other organs
* severe chronic extrahepatic disease including chronic obstructive pulmonary disease combined with respiratory failure, coronary heart disease with cardiac function level 3 (NYHA), myocardial infarction in the 3 months before admission, diabetes with severe complications and chronic kidney disease with end-stage renal failure
* receiving immunosuppressive drugs for reasons other than chronic liver disease

Ages: 15 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: chronic liver disease patients（having liver dysfunction more than 6 months） with acute liver injury[having ALT(alanine aminotransferase)>3NL(normal level),AST(aspartate aminotransferase)>3NL or TB(total bilirubin)>2NL within 1 week before enrollment] or acute decompensation[having ascites, hepatic encephalopathy, bacterial infection ,gastrointestinal bleeding or jaundice(TB>5NL)within 1 month before enrollment].
Sampling Method: Probability Sample
Enrollment: 2600 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hai Li, Study Director — RenJi Hospital
Locations (16):
- China (16):
  - Ditan Hospital of integrated traditional Chinese and Western Medicine Center, Beijing, Beijing Municipality
  - Southwest Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Fuzhou general hospital of Xiamen university, Fuzhou, Fujian
  - Southern hospital infection department, Guangzhou, Guangdong
  - Affiliated Hospital of the Armed Police Logistics College, Tianjingcun, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Wuhan Union Hospital of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Fudan University Huashan hospital, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan hospital, Shanghai, Shanghai Municipality
  - Renji hospital of Shanghai Jiao Tong University School of Medical, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohnishi H, Sugihara J, Moriwaki H, Muto Y. [Acute-on-chronic liver failure]. Ryoikibetsu Shokogun Shirizu. 1995;(7):217-9. No abstract available. Japanese. PMID 8749457
- [Background] Kim TY, Kim DJ. Acute-on-chronic liver failure. Clin Mol Hepatol. 2013 Dec;19(4):349-59. doi: 10.3350/cmh.2013.19.4.349. Epub 2013 Dec 28. PMID 24459638
- [Background] Olson JC, Wendon JA, Kramer DJ, Arroyo V, Jalan R, Garcia-Tsao G, Kamath PS. Intensive care of the patient with cirrhosis. Hepatology. 2011 Nov;54(5):1864-72. doi: 10.1002/hep.24622. PMID 21898477
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Background] Jalan R, Saliba F, Pavesi M, Amoros A, Moreau R, Gines P, Levesque E, Durand F, Angeli P, Caraceni P, Hopf C, Alessandria C, Rodriguez E, Solis-Munoz P, Laleman W, Trebicka J, Zeuzem S, Gustot T, Mookerjee R, Elkrief L, Soriano G, Cordoba J, Morando F, Gerbes A, Agarwal B, Samuel D, Bernardi M, Arroyo V; CANONIC study investigators of the EASL-CLIF Consortium. Development and validation of a prognostic score to predict mortality in patients with acute-on-chronic liver failure. J Hepatol. 2014 Nov;61(5):1038-47. doi: 10.1016/j.jhep.2014.06.012. Epub 2014 Jun 17. PMID 24950482
- [Background] Sun QF, Ding JG, Xu DZ, Chen YP, Hong L, Ye ZY, Zheng MH, Fu RQ, Wu JG, Du QW, Chen W, Wang XF, Sheng JF. Prediction of the prognosis of patients with acute-on-chronic hepatitis B liver failure using the model for end-stage liver disease scoring system and a novel logistic regression model. J Viral Hepat. 2009 Jul;16(7):464-70. doi: 10.1111/j.1365-2893.2008.01046.x. Epub 2009 Apr 29. PMID 19413694
- [Background] Gines P, Schrier RW. Renal failure in cirrhosis. N Engl J Med. 2009 Sep 24;361(13):1279-90. doi: 10.1056/NEJMra0809139. No abstract available. PMID 19776409
- [Background] Blei AT, Cordoba J; Practice Parameters Committee of the American College of Gastroenterology. Hepatic Encephalopathy. Am J Gastroenterol. 2001 Jul;96(7):1968-76. doi: 10.1111/j.1572-0241.2001.03964.x. PMID 11467622
- [Background] Wiesner R, Edwards E, Freeman R, Harper A, Kim R, Kamath P, Kremers W, Lake J, Howard T, Merion RM, Wolfe RA, Krom R; United Network for Organ Sharing Liver Disease Severity Score Committee. Model for end-stage liver disease (MELD) and allocation of donor livers. Gastroenterology. 2003 Jan;124(1):91-6. doi: 10.1053/gast.2003.50016. PMID 12512033
- [Background] Bajaj JS, O'Leary JG, Reddy KR, Wong F, Olson JC, Subramanian RM, Brown G, Noble NA, Thacker LR, Kamath PS; NACSELD. Second infections independently increase mortality in hospitalized patients with cirrhosis: the North American consortium for the study of end-stage liver disease (NACSELD) experience. Hepatology. 2012 Dec;56(6):2328-35. doi: 10.1002/hep.25947. PMID 22806618
- [Result] Gu WY, Xu BY, Zheng X, Chen J, Wang XB, Huang Y, Gao YH, Meng ZJ, Qian ZP, Liu F, Lu XB, Shang J, Li H, Wang SY, Sun X, Li H. Acute-on-Chronic Liver Failure in China: Rationale for Developing a Patient Registry and Baseline Characteristics. Am J Epidemiol. 2018 Sep 1;187(9):1829-1839. doi: 10.1093/aje/kwy083. PMID 29762630
- [Derived] Zhang Y, Tan W, Wang X, Zheng X, Huang Y, Li B, Meng Z, Gao Y, Qian Z, Liu F, Lu X, Shi Y, Shang J, Yan H, Zheng Y, Zhang W, Gu W, Qiao L, Deng G, Zhou Y, Hou Y, Zhang Q, Xiong S, Liu J, Duan L, Chen R, Chen J, Jiang X, Luo S, Chen Y, Jiang C, Zhao J, Ji L, Mei X, Li J, Li T, Zheng R, Zhou X, Ren H, Cheng X, Guo L, Li H; Chinese (Acute on) Chronic Liver Failure Consortium (Ch-CLIF.C). Metabolic biomarkers significantly enhance the prediction of HBV-related ACLF occurrence and outcomes. J Hepatol. 2023 Nov;79(5):1159-1171. doi: 10.1016/j.jhep.2023.07.011. Epub 2023 Jul 29. PMID 37517452
- [Derived] Wang T, Tan W, Wang X, Zheng X, Huang Y, Li B, Meng Z, Gao Y, Qian Z, Liu F, Lu X, Yan H, Zheng Y, Zhang W, Yin S, Gu W, Zhang Y, Dong F, Wei J, Deng G, Xiang X, Zhou Y, Hou Y, Zhang Q, Xiong S, Liu J, Long L, Chen R, Chen J, Jiang X, Luo S, Chen Y, Jiang C, Zhao J, Ji L, Mei X, Li J, Li T, Zheng R, Zhou X, Ren H, Shi Y, Li H; Chinese (Acute on) Chronic Liver Failure Consortium (Ch-CLIF.C). Role of precipitants in transition of acute decompensation to acute-on-chronic liver failure in patients with HBV-related cirrhosis. JHEP Rep. 2022 Jul 5;4(10):100529. doi: 10.1016/j.jhepr.2022.100529. eCollection 2022 Oct. PMID 36052222
- [Derived] Mei X, Li H, Deng G, Wang X, Zheng X, Huang Y, Chen J, Meng Z, Gao Y, Liu F, Lu X, Shi Y, Zheng Y, Yan H, Zhang W, Qiao L, Gu W, Zhang Y, Xiang X, Zhou Y, Sun S, Hou Y, Zhang Q, Xiong Y, Zou C, Chen J, Huang Z, Li B, Jiang X, Zhong G, Wang H, Chen Y, Luo S, Gao N, Liu C, Li J, Li T, Zheng R, Zhou X, Ren H, Yuan W, Qian Z. Prevalence and clinical significance of serum sodium variability in patients with acute-on-chronic liver diseases: a prospective multicenter study in China. Hepatol Int. 2022 Feb;16(1):183-194. doi: 10.1007/s12072-021-10282-8. Epub 2022 Jan 17. PMID 35037228
- [Derived] Sun S, Xu B, Tan W, Xiang X, Zhou Y, Dan Y, Guo Y, Tan Z, Deng G. Testosterone and Estradiol as Novel Prognostic Indicators for HBV-Related Acute-on-Chronic Liver Failure. Front Med (Lausanne). 2021 Sep 8;8:729030. doi: 10.3389/fmed.2021.729030. eCollection 2021. PMID 34568387
- [Derived] Ouyang R, Li H, Xia J, Wang X, Zheng X, Huang Y, Meng Z, Gao Y, Qian Z, Liu F, Lu X, Shi Y, Shang J, Liu J, Deng G, Zheng Y, Yan H, Zhang W, Qiao L, Jiang X, Wang H, Zhong G, Li B, Chen J. Lower platelet counts were associated with 90-day adverse outcomes in acute-on-chronic liver disease patients. Ann Palliat Med. 2021 Sep;10(9):9342-9353. doi: 10.21037/apm-21-1019. Epub 2021 Aug 13. PMID 34412498
- [Derived] Chen J, Huang ZB, Li H, Zheng X, Chen JJ, Wang XB, Qian ZP, Liu XX, Fan XG, Hu XW, Liao CJ, Long LY, Huang Y. Early Diagnostic Biomarkers of Sepsis for Patients with Acute-on-Chronic Liver Failure: A Multicenter Study. Infect Dis Ther. 2021 Mar;10(1):281-290. doi: 10.1007/s40121-020-00362-x. Epub 2020 Nov 4. PMID 33146854
- [Derived] Li B, Gao Y, Wang X, Qian Z, Meng Z, Huang Y, Deng G, Lu X, Liu F, Zheng X, Li H, Chen J. Clinical features and outcomes of bacterascites in cirrhotic patients: A retrospective, multicentre study. Liver Int. 2020 Jun;40(6):1447-1456. doi: 10.1111/liv.14418. Epub 2020 Mar 17. PMID 32128975
- [Derived] Zhang Y, Xu BY, Wang XB, Zheng X, Huang Y, Chen J, Meng ZJ, Gao YH, Qian ZP, Liu F, Lu XB, Shi Y, Shang J, Li H, Wang SY, Yin S, Sun SN, Hou YX, Xiong Y, Chen J, Li BL, Lei Q, Gao N, Ji LJ, Li J, Jie FR, Zhao RH, Liu JP, Lin TF, Chen LY, Tan WT, Zhang Q, Zou CC, Huang ZB, Jiang XH, Luo S, Liu CY, Zhang YY, Li T, Ren HT, Wang SJ, Deng GH, Xiong SE, Liu XX, Wang C, Yuan W, Gu WY, Qiao L, Wang TY, Wu DD, Dong FC, Li H, Hua J. Prevalence and Clinical Significance of Portal Vein Thrombosis in Patients With Cirrhosis and Acute Decompensation. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2564-2572.e1. doi: 10.1016/j.cgh.2020.02.037. Epub 2020 Feb 25. PMID 32109631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only INPATIENTS who met inclusion criteria were recruited.
Pre-assignment Details: Did not meet inclusion criteria (n = 1,306) ;Age <15 years or ≥80 years (n = 36);Pregnant (n = 22);Liver malignancies (n = 514);Malignancies in other organs (n = 77);Severe chronic extrahepatic disease (n = 107);Received immunosuppressive drugs for reasons other than chronic liver disease (n = 21);Withdrew informed consent (n = 73);Other (n = 205)
Groups:
- Acute-on-Chronic Liver Disease Inpatients: 1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients and non-alcoholic fatty liver disease patients,.
  2. ALI(acute liver injury): including [ALT>3NL(normal level),AST>3NL or TB>2NL within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy, bacterial infection, gastrointestinal bleeding or jaundice(TB>5NL) within 1 month before enrollment)]
  3. Standary therapy for chronic liver disease with ATI and/or AD
Period: Recruitment
Arm/Group | Acute-on-Chronic Liver Disease Inpatients
Started | 2600 (2600 is the number of inpatients who met our eligibility.)
Completed | 2600 (2361 patients were excluded according to our exclusion criteria,2600 patients remained.)
Not Completed | 0
Period: 28-Days Hospitalization and Observation
Arm/Group | Acute-on-Chronic Liver Disease Inpatients
Started | 2600
Liver Transplantation | 124
Death | 74
Completed | 2600 (Death and receiving Liver transplantation are two end points of our observation.)
Not Completed | 0
Period: Clinic or Telephone Follow-up
Arm/Group | Acute-on-Chronic Liver Disease Inpatients
Started | 2600
One-year Liver Transplantation | 182
One-year Death | 475
Completed | 2529
Not Completed | 71
Not completed — Lost to Follow-up | 71

BASELINE CHARACTERISTICS:
Groups:
- Acute-on-Chronic Liver Disease Inpatients: 1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients and non-alcoholic fatty liver disease patients.
  2. ALI(acute liver injury): including [ALT>3NL(normal level),AST>3NL or TB>2NL within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy, bacterial infection, gastrointestinal bleeding or jaundice(TB>5NL) within 1 month before enrollment)].
  3. Standary therapy for chronic liver disease with ATI and/or AD.
Arm/Group | Acute-on-Chronic Liver Disease Inpatients
Number analyzed (Participants) | 2600
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.34 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 685
  Male | 1915
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2600
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 2600
Etiology（Related to HBV） [Count of Participants; unit: Participants]
  Related to HBV | 1859
  Not related to HBV | 741
blood routine test [Mean (Standard Deviation); unit: cell *10^9/L] — blood routine test(WBC and Platelet)
  cell *10^9/L
    White blood cell | 5.90 (4.64)
    Platelet | 109 (78)
INR [Mean (Standard Deviation); unit: ratio] — international normalized ratio
  ratio | 1.64 (0.78)
Other Liver Biochemical Parameters [Mean (Standard Deviation); unit: U/L] — other biochemical parameters of liver function from patients' blood sample
  U/L
    Alanine aminotransferase | 328.21 (515.93)
    Aspartate aminotransferase | 262.07 (98.69)
    γ-Glutamyltransferase | 127.78 (182.83)
    Alkaline phosphatase | 153.13 (126.70)
Biochemical Parameters [Mean (Standard Deviation); unit: mg/dL] — basic biochemical parameters of blood sample
  mg/dL
    Serum bilirubin | 9.30 (10.32)
    Serum creatinine | 0.87 (0.63)
Serum sodium [Mean (Standard Deviation); unit: mmol/L] — Serum sodium from blood sample
  mmol/L | 137.38 (5.94)

OUTCOME MEASURES:

1. Primary Outcome: 28-day Mortality,28-day Liver-transplantation Free Mortality& 28-day Liver Transplantation Rate
Description: liver-transplantation free mortality refers to number of participants who died in the absence of receiving a liver transplant divided by number of participants without liver transplant.
Time Frame: up to 28 days
Population: liver-transplantation free mortality refers to number of participants who died in the absence of receiving a liver transplant divided by liver-transplantation free participants
Measure: Count of Participants; unit: Participants
Groups:
- Acute-on-Chronic Liver Disease: 1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients and non-alcoholic fatty liver disease patients,.
  2. ALI(acute liver injury): including [ALT>3NL(normal level),AST>3NL or TB>2NL within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy, bacterial infection, gastrointestinal bleeding or jaundice(TB>5NL) within 1 month before enrollment)]
  3. Standary therapy for chronic liver disease with ATI and/or AD
Arm/Group | Acute-on-Chronic Liver Disease
Number analyzed (Participants) | 2600
Participants
  28-day Mortality | 74
  28-day Liver Transplantation Rate at 28 days | 124
  28-day liver transplantation free mortality: number analyzed (Participants) | 2476
  28-day liver transplantation free mortality | 74

2. Secondary Outcome: 90-day Mortality Rates, 90-day Liver Transplantation Free Mortality and Liver Transplantation Rate
Description: as for outcome 1
Time Frame: up to 90 days
Population: Mortality will be respectively calculated together with the liver transplantation rate (as the rate of ''incidence'')and independently (as the ''liver transplantation free mortality'') respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute-on-Chronic Liver Disease Inpatients
Number analyzed (Participants) | 2600
Participants
  90-day mortality rate | 333
  90-day liver transplantation rate | 171
  90-day liver transplantation free mortality: number analyzed (Participants) | 2429
  90-day liver transplantation free mortality | 333

3. Secondary Outcome: 180-day Mortality Rate and Liver Transplantation Rate
Description: Mortality will be respectively calculated together with the liver transplantation rate (as the rate of ''incidence'')and independently (as the ''liver transplantation free mortality'') respectively.
Time Frame: up to 180 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acute-on-Chronic Liver Disease Inpatients
Number analyzed (Participants) | 2600
Participants
  180-day mortality rate | 403
  180-day liver transplantation rate | 177
  180-day liver transplantation free mortality': number analyzed (Participants) | 2423
  180-day liver transplantation free mortality' | 403

4. Other Pre Specified Outcome: The Appearance and Number of Organ Failure
Description: The appearance and number of organ failure（including liver, coagulation, renal, circulation, brain, respiratory system） will be evaluated and reported at 1, 4, 7, 14, 21 and 28 days (or last visit)during patients' hospitalization.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Acute-on-Chronic Liver Disease
Number analyzed (Participants) | 2600
Participants | 261

5. Other Pre Specified Outcome: Models for Disease Severity
Description: MELD score, MELD-Na score, CLIF-SOFA score, SOFA score and APACHE scores will be calculated and reported at 1, 4, 7, 14, 21 and 28 days (or last visit) during patients' hospitalization.
  MELD：Model for end-stage liver disease MELD-Na： Model for end-stage liver disease - sodium SOFA：sequential organ failure assessment CLIF-SOFA：chronic liver failure-sequential organ failure assessment APACHE：Acute Physiology And Chronic Health Evaluation
Time Frame: Up to 28 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Serum Bilirubin
Description: be collected and reported at 28 or last visit before discharge
Time Frame: Up to 28 days
Population: participants who had TB analysis at 28 day after administration
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Acute-on-Chronic Liver Disease
Number analyzed (Participants) | 1011
mg/dL | 9.3 (10.32)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Acute-on-Chronic Liver Disease: 1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients; and non-alcoholic fatty liver disease patients.
  2. ALI(acute liver injury): including [ALT>3NL(normal level),AST>3NL or TB>2NL within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy, bacterial infection gastrointestinal bleeding or jaundice(TB>5NL)within 1 month before enrollment)].
  3. Standary therapy
Arm/Group | Acute-on-Chronic Liver Disease
All-Cause Mortality (participants affected / at risk) | 475/2600
Serious Adverse Events (participants affected / at risk) | 0/2600
Other Adverse Events (participants affected / at risk) | 0/2600

LIMITATIONS AND CAVEATS:
1. ACLF has no pathological criteria yet thus the diagnosis is made based on clinical data and mortality.
2. The diagnosis of cirrhosis was based on both clinical data and imaging instead of liver biopsy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02457637/Prot_SAP_000.pdf
  • Informed Consent Form (2014-11-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT02457637/ICF_001.pdf